CLINICAL TRIAL: NCT01711099
Title: Hungarian Study on the Efficacy of Extracorporeal Shockwave Myocardial Revascularization in Patients With Therapy-refracter Angina Pectoris
Brief Title: Efficacy of Extracorporeal Shockwave Myocardial Revascularization
Acronym: ANGEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salus Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANGEL_v01
Record Dates: First submitted 2012-10-16; First posted 2012-10-22 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Refractory Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Therapeutics

ARMS (1):
- ESMR treated (Experimental)
  Interventions: Device: device for Extracorporeal Shockwave Myocardial Revascularization (ESMR) therapy

INTERVENTIONS:
Device: device for Extracorporeal Shockwave Myocardial Revascularization (ESMR) therapy
  Other Names: Cardiospec system

SUMMARY:
Clinical research to justify effectiveness of the Extracorporeal Shockwave Myocardial Revascularization (ESMR) Therapy for treatment of patients with reversible myocardial ischemia secondary to Coronary Artery Disease (CAD) and therapy resistant stable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a signed Informed Consent Form.
* Patient's current and past medical condition and status be assessed using previous medical history, complete physical examination and the physicians (principle investigator's) medical opinion.
* Patient is diagnosed with chronic angina pectoris for at least 6 weeks. Diagnosis is based on medical history, complete physical examination, and core labs.
* Patients who no longer receive benefit from additional revascularization procedures (i.e. CABG or Angioplasty). Certification will be made by Heart Team.
* Patient demonstrates Exercise Tolerance Time (ETT) duration < 10 minutes on Modified Bruce protocol.
* Patient had at least one documented myocardial segment with reversible ischemia.
* Patient is under optimum medical therapy for angina for at least 6 weeks. The optimal treatment plan is tailored to a person's age, the presence of other medical conditions, lifestyle, medication side effects, etc. Medical therapies for stable angina include ACE-inhibitors, Nitrates, Beta Blockers and Calcium Channel Blockers, trimetazidine, ivabradin. Combination of any of 3 above mentioned drugs will be considered as optimum medical therapy.
* Patient has an echocardiographic acoustic window to the target area in the myocardium utilizing one of the following views: apical 2 chamber view (2CH), apical 4 chamber view (4CH), modified parasternal long axis view (LAX) and parasternal short axis view (SAX).

Exclusion Criteria:

* Patient who will substantially benefit from additional revascularization procedures such as additional CABG or angioplasty therapies. This determination will be made and certified by the Heart Team.
* Patient has active endocarditis, myocarditis or pericarditis.
* Patient with moderately severe or severe valvular disease.
* Patient with known intraventricular thrombus.
* Patients who have active or non-active implantables, such as pacemakers, defibrillators, abandoned leads, or electrodes.
* Patient for who shock waves applied over any implanted device that releases substances or medications to the periphery (such as insulin pumps).
* Patient is pregnant.
* Patient with severe chronic lung disease (emphysema, pulmonary fibrosis) with difficult access to ultrasonic acoustic window.
* Patients for who shock waves applied over the area of healing fracture.
* Patients for who shock waves applied over the area of bone growth.
* Patients for who shock waves applied to the area of malignancy.
* Prior invasive malignancy, except non-melanomatous skin cancer or other malignancies with a documented disease-free survival for a minimum of 5 years.
* By the physician decision there is underlying concomitant disease or circumstance what may negatively influence the management of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in myocardial ischaemia profile during dobutamine induced stress echocardiography | baseline and 6 months

SECONDARY OUTCOMES:
Improvement in the angina pectoris CCS Stage | baseline and 3, 6 months
Improvement in angina status using Seattle Angina Questionnaire | baseline and 3, 6 months
The change in walking time using the modified Bruce exercise test | baseline and 3, 6 months
The change in basal transthoracal echocardiographic parameters | baseline and 3, 6 months
The decrease in nitrate use during the unchanged everyday activity reported by the patients in the "Nitrate Usage Log" | baseline and 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Béla Merkely, Prof, Principal Investigator — Semmelweis University Heart Center
Locations (2):
- Hungary (2):
  - Kelen Hospital, Budapest
  - Semmelweis University Heart Center, Budapest